CLINICAL TRIAL: NCT01895907
Title: SCOPE and Special Olympics
Acronym: SCOPE/SO
Status: Completed | Type: Observational
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Other Study IDs: 15528
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2013-07

CONDITIONS: Special Olympic Athletes' Life Participation
Keywords: Special Olympics; occupational therapy; SCOPE; life participation improvement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Special Olympic athletes

SUMMARY:
The purpose of this study is to examine if Special Olympic athletes's life participation improves through involvement with Special Olympics. This project will be undertaken in coordination with Special Olympics entities from Texas and around the nation to determine how involvement in Special Olympics improves the strengths and limitations of their athletes. The Short Child Occupational Profile (SCOPE) will be used to gather this information from the parents and coaches. The SCOPE measures the impact that personal and environmental factors have on a child or youth's occupational participation.

DETAILED DESCRIPTION:
The research team members will not have contact with the Special Olympic athletes. Parents and coaches will be the only individuals who have contact with the athletes. Participants will be assured that their participation is completely voluntary. If they agree to participate in the research an informed assest form will be explained by a parent, guardian, or coach and they will be asked to sign it. Parents will be asked to sign a consent form for their child's participation in the study. Coaches will administer the SCOPE as a pre/post-test outcome measure. Parents will submit the Parent form of the SCOPE and the coaches will submit the SCOPE Clinical Data Summary Form. All data will be de-identified and sent in form the coaches. The TWU special olympics research team will compile de-identified data from a pre-test and post-test utilizing the SCOPE. A codebook that links the ID number with the participants will be kept by the coaches. The research team may be able to trace assented data collected through the TWU data collection protocol back to the coaches. Participating athletes will not be contacted by the PI and no contact information will be collected. In the case of an unexpected or adverse event, or if the participants request to be contacted, attempts may be made to find the subjects contact information through the coaches. De-identified data collected by the TWU Special Olympic research team or other Key Research personnel will be stored on a password protected computer or in a locked file cabinet in a locked office in the department of occupational therapy at Texas Woman's University in Houston. The raw data collected will not be made available to anyone other than the PI and immediate study research personnel. Data is entered into the database using the ID number, and the computer database is password protected. The raw data is not going to be shared. The data will be kept in a locked file cabinet within the research office of the databases destroyed 4 years after the end of the study. The results of the analysis, which may include information from the data, will be kept on a password secure computer indefinitely. The data collected from pre-tests and post-tests will then be compiled and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* new members (within 2 years),
* English-speaking,
* U.S. citizens, and
* must be 7 years or older at the time of assess.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participating athletes will be recruited through the coaches. Participants recruited under the TWU collection protocol will be informed that they are being asked to be a subject in a research study to determine if there is a change in levels of participation in other areas of life for athletes involved in special olympics.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Short Child Occupational Profile | up to 3 years-estimated
  To determine if there is a change in levels of participation in other areas of life for athletes involved in Special Olympics

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Bowyer, EdD, OTR, BCN, FAOTA, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Houston, Texas, United States